CLINICAL TRIAL: NCT03539250
Title: Dose Constraints for the Temporal Lobes During the Optimization of Intensity-modulated Radiotherapy Treatment Plans for Nasopharyngeal Carcinoma
Brief Title: Dose Constraints for the Temporal Lobes of Intensity-modulated Radiotherapy Treatment Plans for Nasopharyngeal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qiang Xu, head of Science and Euducation Division, Jiangxi Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zl2017
Record Dates: First submitted 2018-03-10; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Injury; Temporal Region
Keywords: Radiation-induced temporal lobe injury;NPC; Nasopharyngeal carcinoma; Intensity-modulated radiotherapy
MeSH Terms: conditions — Wounds and Injuries; Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMRT with and without chemotherapy (Experimental): Subdivision of the PTVnx into regions with different prescribed absorbed doses (PTVsv1,PTVsv2, PTVsv2 is the overlaps between PTVnx and temporal lobe) can be used in cases for which the PTVnx overlaps temporal lobe. When the volume of PTVsv2 is less than 0.2 cubic centimeter (cc), the prescribe dose for PTVsv2 is as the same as that of the PTVsv1, D1cc 63.1Gy, Dmax 72.9Gy for TL (32 fractions). When the volume of PTVsv2 is between 0.2 cc and 0.5cc, the prescribe dose for PTVsv2 is 66Gy, D1cc 63.1Gy, Dmax 72.9Gy for TL (32 fractions). When the volume of PTVsv2 is between 0.5 cc and 1cc, the prescribe dose for PTVsv2 is 66Gy, D1cc 65.8Gy, Dmax 75.2Gy for TL (32 fractions).
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: IMRT — IMRT with and without chemotherapy

SUMMARY:
Radiation-induced temporal lobe injury (TLI) is usually devastating to patients; however, there is a poor understanding of TLI in nasopharyngeal carcinoma (NPC) patients treated with IMRT. Knowledge of the dose tolerance of the TL is essential, in order to predict the safety of intensity-modulated radiotherapy (IMRT) treatment plans. In our previous studies, D1cc (the dose to 1ml of the TL volume) and Dmax (the maximum point dose) were the significant predictors of TLI development. The purpose of this study is to evaluate the feasibility of dose constraints based on D1cc and Dmax for the temporal lobes following IMRT for NPC.

DETAILED DESCRIPTION:
The prescribe dose was 66-70Gy to the PTV of the GTVnx, 60Gy to the PTV of CTV1(i.e., high-risk regions),54-56Gy to the PTV of CTV2(i.e., low-risk regions),and 64-66Gy to the PTV of the GTVnd for the metastatic cervical lymph nodes in 30-33 fractions. For the GTV and CTV, the target volumes that received more than 95% of the prescribed dose was used to reflect the target coverage. Subdivision of the PTVnx into regions with different prescribed absorbed doses (PTVsv1,PTVsv2, PTVsv2 is the overlaps between PTVnx and temporal lobe) can be used in cases for which the PTVnx overlaps temporal lobe. When the volume of PTVsv2 is less than 0.2 cubic centimeter (cc), the prescribe dose for PTVsv2 is as the same as that of the PTVsv1, D1cc 63.1Gy, Dmax 72.9Gy for TL (32 fractions). When the volume of PTVsv2 is between 0.2 cc and 0.5cc, the prescribe dose for PTVsv2 is 66Gy, D1cc 63.1Gy, Dmax 72.9Gy for TL (32 fractions). When the volume of PTVsv2 is between 0.5 cc and 1cc, the prescribe dose for PTVsv2 is 66Gy, D1cc 65.8Gy, Dmax 75.2Gy for TL (32 fractions).

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed and confirmed histopathologic diagnosis of nasopharyngeal squamous cell carcinoma, types WHO II-III, Stage I-IVA (AJCC staging, 2017, 8th edition), treated with intensity-modulated radiotherapy.
* No head and neck surgery of the primary tumor or lymph nodes except for incisional or excisional biopsies.
* Age between 18 years and 70 years.
* Karnofsky score ≥80
* WBC≥ 4,000/ul, platelets≥ 100,000/ul; serum creatinine≤ 1.6 mg/dl or 24hr. calculated creatinine clearance ≥ 60ml/min.
* Must undergo pre-treatment evaluation of tumor extent and tumor measurement. Tumor may be measurable or evaluable.
* Signed study-specific consent form prior to study entry.

Exclusion Criteria:

* Stage IVB
* Evidence of distant metastases
* Previous irradiation for head and neck tumor ≤ 6 months prior to study entry
* Previous chemotherapy ≤ 6 months prior to study entry
* Patient is on other experimental therapeutic cancer treatment
* Other malignancy except non-melanoma skin cancer or a carcinoma not of head and neck origin and controlled at least 5 years
* Active untreated infection
* Major medical or psychiatric illness, which in the investigator's opinions, would interfere with either the completion of therapy and follow-up or with full and complete understanding of the risks and potential complications of the therapy
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2018-06-10 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of radiation-induced temporal lobe injury at 5 years | 5 years
  The incidence of radiation-induced temporal lobe injury at 5 years will be calculated

SECONDARY OUTCOMES:
Local recurrence-free survival at 5 years | 5 years
  Local recurrence-free survival at 5 years will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Gao Li, MD, Principal Investigator — Jiangxi cancer hospital, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT03539250/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT03539250/ICF_001.pdf